CLINICAL TRIAL: NCT02370290
Title: CT Metrology: Quantitative Imaging Metrics With Advanced Visualization Tools for Cancer Imaging
Brief Title: Quantitative Imaging Metrics From CECT in Measuring Disease Response or Progression in Patients With Kidney Cancer
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 4K-13-2; NCI-2014-02547 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HS-13-00256; 4K-13-2 (Other: USC Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2015-02-17; First posted 2015-02-24 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational (QIM): Patients' clinical and imaging data are collected from routine multiphase CECT imaging and used to establish and validate the classification/prediction rule for QIM.
  Interventions: Other: Medical Chart Review; Other: Informational Intervention

INTERVENTIONS:
Other: Medical Chart Review — Clinical and imaging information collected
  Other Names: Chart Review
Other: Informational Intervention — Clinical and imaging data collected

SUMMARY:
This pilot research trial studies quantitative imaging metrics derived from contrast enhanced computed tomography (CECT) in enhancing assessment of disease status in patients with kidney cancer. Quantitative imaging is the extraction of quantifiable features from radiological images for the assessment of disease status. Collecting quantitative imaging metrics from CECT imaging may help doctors predict tumor aggressiveness and nuclear grade (tumor stage) and assess treatment response and prognosis in cancer imaging.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate the role of quantitative imaging metrics (QIM) as a potential DIAGNOSTIC biomarker.

II. To investigate if QIM parameters can differentiate clear cell renal cell carcinoma (RCC) from papillary RCC.

III. To evaluate the tumor grade of the target lesion as assessed by QIM from CECT for agreement with the pathological (Fuhrman) grade.

IV. To investigate the role of QIM as a potential PROGNOSTIC biomarker. V. To develop a novel method of calculating renal tumor contact surface area (CSA) using advanced image-processing technology (MATLAB®, 3 dimension [D] Synapse) and predict peri-operative variables such as blood loss, operative time and post-operative estimated glomerular filtration rate (eGFR) in patients undergoing partial nephrectomy (PN).

VI. To develop QIM that would help in predicting postoperative functional outcomes such as predicted surgically resected volume and postoperative glomerular filtration rate (GFR).

OUTLINE:

Patients' clinical and imaging data are collected from routine multiphase CECT imaging and used to establish and validate the classification/prediction rule for QIM.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a renal mass who are scheduled for surgery for presumed RCC
* Subjects scheduled for standard of care contrast enhanced CT examination at USC Norris Comprehensive Cancer Center
* Subjects competent to sign study specific written informed consent

Exclusion Criteria:

* Subjects who are pregnant
* Subjects who cannot consent for themselves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients' clinical and imaging data from the University of Southern California/Norris Comprehensive Cancer Center and Keck Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Agreement between QIM predicted and pathologically determined tumor class (clear cell renal cell carcinoma [ccRCC] vs papillary [p]RCC) | Baseline
  Cohen's kappa coefficient will be used to examine the agreement between QIM predicted and pathologically determined tumor class (ccRCC vs. pRCC).
Agreement between QIM predicted and pathologically determined tumor (Fuhrman) grade | Baseline
  Examined using weighted kappa coefficient.
Agreement between QIM predicted and clinically observed perioperative measurements such as blood loss, operative time, and eGFR | Baseline
  Examined using two-way random single measure with absolute agreement.
Agreement between QIM predicted and clinical determined postoperative eGFR | Baseline
  Examined using two-way random single measure with absolute agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Duddalwar, Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States